CLINICAL TRIAL: NCT00447850
Title: Endometrial Gene Expression Profile in Controlled Ovarian Stimulation Cycles With Premature Luteinization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Responsible Party: Dr. Elena Labarta, Instituto Valenciano de Infertilidad
Other Study IDs: VLC-EL-1006- 307-2
Record Dates: First submitted 2007-03-13; First posted 2007-03-15 (Estimated); Last update posted 2009-09-21 (Estimated); Status verified 2009-09

CONDITIONS: Premature Luteinization

INTERVENTIONS:
Procedure: endometrial biopsy

SUMMARY:
Previous studies have suggested that premature luteinization (PL)during controlled ovarian stimulation (COS) decreases the implantation rate due to a negative effect on the endometrium receptivity. This study aims to describe the impact on endometrial gene expression of PL in GnRH antagonist and GnRH agonist cycles.

ELIGIBILITY:
Inclusion Criteria:

* Oocyte donors
* Age between 18-35 years old
* BMI 18-29
* NORMOGONADOTROPHICS
* PROGESTERONE ≥ 1.2 ng/ml on hCG day

Exclusion Criteria:

* PolyCystic Ovarian Syndrome (PCOS)
* Endometriosis

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2007-04; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elena Labarta, MD, Principal Investigator — Instituto Valenciano de la Infertilidad
Locations (1):
- Ivi Valencia, Valencia, Spain